CLINICAL TRIAL: NCT02878122
Title: Study of Predictive Factors of Chemoresistance in Ovarian Cancer
Acronym: FaCliBioCCo
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC15_3007_FaCliBioCCo
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; chemo resistance; predictive factors; cohort study; bio bank
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Antineoplastic Protocols; CP protocol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — surgical sampling, blood plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with epithelial ovarian cancer: Cancer treatment
  Interventions: Procedure: Cancer treatment

INTERVENTIONS:
Procedure: Cancer treatment — Chemotherapy and laparoscopic surgery
  Other Names: Carboplatin, Taxol

SUMMARY:
Epithelial ovarian cancer (EOC) has a poor prognosis. EOC management requires debulking surgery and chemotherapy based on taxol and carboplatine. Initial response is often good, but most often a recurrence occurred in the first 18 months. Early recurrence signs chemoresistance and palliative treatment. The study of predictive clinical or biological factors is required to adapt therapeutic and develop new treatments.

ELIGIBILITY:
Inclusion Criteria:

* patient > 18 years of age
* patient with histological proven epithelial ovarian cancer

Exclusion Criteria:

* patients who can not give their own consent
* patients without ovarian cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epithelial ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-03; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Chemoresistance defined by clinical recurrence | 6 months after the end of chemotherapy
Chemoresistance defined by biological recurrence | 6 months after the end of chemotherapy
Chemoresistance defined by radiological recurrence | 6 months after the end of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: LAVOUE Vincent, Pr, Principal Investigator — Rennes University Hospital
Locations (1):
- LAVOUE, Rennes, France

IPD SHARING:
Plan to Share IPD: No